CLINICAL TRIAL: NCT06412432
Title: Exercise Training and Rehabilitation In Cardiac Amyloidosis: ERICA-Study
Brief Title: Exercise Training and Rehabilitation In Cardiac Amyloidosis
Acronym: ERICA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alberto Maria Marra, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERICA562023CRCA
Record Dates: First submitted 2024-04-15; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac Amyloidosis; wild-type transthyretin; Exercise Training; Rehabilitation; Cardiomyopathies; Heart Failure
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Cardiomyopathies; Heart Failure | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients enrolled will be handled in the outpatient's clinic of Cardiometabolic Rehabilitation Program of the Federico II University Hospital of Naples for exercise training and cardiac rehabilitation intervention. Patients will be randomized in blocks to two groups. Specifically, the primary intervention (ET-1) and the control group who won't undergo exercise training (No-ET). Following baseline assessments of both groups at baseline, the ET-1 group will be subjected to exercise training program of 2 weekly sessions for 12 weeks. After 12 weeks, both groups will be reassessed and patients belonging to group No-ET will be offered to undergo the same ET program for further 12 weeks. Those who will accept will join the secondary training group (ET-2). Primary endpoint will be the distance obtained at the 6-minute walk test (6MWD) performed at baseline and after 12-weeks of treatment in pooled ET-1 and ET-2 groups compared to No-ET.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Patients will undergo exercise training, nutritional advice, smoking cessation, lipid profile evaluation, control and management of body weight and abdominal circumference; evaluation of the drug therapy in progress; psycho-social evaluation.
  Interventions: Other: Exercise training (ET1+ET2)
- Controls (Active Comparator): control group who won't undergo exercise training and will be managed with optimal medical therapy
  Interventions: Behavioral: Optimal Medical Therapy (No-ET)

INTERVENTIONS:
Other: Exercise training (ET1+ET2) — Exercise training will consist of continuous aerobic training of moderate intensity on cycle ergometer/treadmill, with a frequency of 2-3 weekly sessions lasting 12 weeks, with exercise intensity of VO2 peak of 40% gradually increasing up to 50-60% of VO2 peak based on individual tolerability and improvement; 55-65% of heart rate at peak; 40-59% of heart rate reserve; 4-6 Metabolic equivalents (METS); the duration of the session will gradually increase from 15-30 min to 45-60 min.
  Arms: Exercise training
Behavioral: Optimal Medical Therapy (No-ET) — Patients will be handled according to optimal medical therapy
  Arms: Controls

SUMMARY:
Notwithstanding the dramatic improvement associated with Tafamidis in Heart Failure (HF) due to wild-type transthyretin cardiac amyloidosis (ATTRwt-CA), remarkable morbidity and mortality still burden this disease. Exercise training (ET) is a first-line recommended treatment for unselected HF patients, whose effects on ATTRwt-CA form remain however unexplored. The investigators hereby present rationale and design of the Exercise training and Rehabilitation in Cardiac Amyloidosis (ERICA) study, whose aim is to determine whether a tailored, supervised ET program might improve exercise capacity in HF due to ATTRwt-CA. This interventional, controlled study will randomize ATTRwt-CA patients into a control group (C) and a primary training group (ET-1). After 12 weeks, patients in group C will be offered to undergo the same ET program (ET-2) for further 12 weeks, considering the last observation as baseline. Primary endpoint will be the distance obtained at the 6-minute walk test (6MWD) performed at baseline and after 12-weeks of treatment in pooled ET-1 and ET-2 groups compared to C. Quality of life, peak oxygen consumption, left and right heart architecture and function, natriuretic peptides will be secondary endpoints. This study will be the first testing the effects of ET in patients with ATTRwt-CA.

DETAILED DESCRIPTION:
Among Systemic amyloidosis, the peculiar deposition of beta-amyloid fibrils agglomerates localized in the interstitial space between the cardiomyocytes characterizes the spectrum of cardiac amyloidosis (AC). All AC phenotypes culminate in a progressive deterioration of cardiac compliance up to a true infiltrative cardiomyopathy with restrictive physiology. Clinical presentation may vary from mildly symptomatic Heart Failure (HF), usually labeled, and mistakenly confused as a classic Heart Failure with preserved ejection fraction (HFpEF) up to a severe scenario of severe cardiac decompensation with fluid overload, marked shortness of breath, fatigue and orthostatic hypotension. Syncope may also appear due to infiltration in the conduction system leading to sinoatrial disease and atrioventricular block. To date, more than 30 proteins responsible for the deposition of fibrils have been identified and of these 9 have been identified as responsible for the cardiac involvement of the disease. AC is determined in 98% of cases by the accumulation of monoclonal light chains of immunoglobulins (AL) or transthyretin (ATTR); the latter can occur either in its hereditary form (ATTRv) or in the wild-type variant (ATTRwt). Although AC is perceived as a rare disease, standing a reported prevalence of around 1/100,000 inhabitants, a recent metanalysis reported AC as underlying HF cause in 13.7% of cases, varying from 15.1% of Heart Failure (HF) with preserved ejection fraction (HFpEF) and 11.3% in reduced fraction phenotype (HFrEF). This mismatch begets the hypothesis that AC is often underdiagnosed, probably due to its challenging diagnosis, the diverse spectrum of clinical presentation ranging from severely compromised clinical cases to rather silent manifestations, and the absence of specific therapies for this condition making until a few years ago AC a true orphan disease. This paradigm has been subverted in recent years, by the emergence of tafamidis, a targeted drug from amyloidosis that binds transthyretin, preventing tetramer dissociation and production of amyloid. Tafamidis has been successfully tested for ATTRwt-AC in a relatively large multicenter, international, double-blind, placebo-controlled, phase 3 trial, the Transthyretin Amyloidosis Cardiomyopathy Clinical Trial (ATTR-ACT), showing a remarkable improvement of the composite outcome of all-cause mortality and hospitalizations due to cardiovascular causes. Apart from Tafamidis, there are no evidence supporting the use of guideline-directed medical therapy (GDMT) used in classical forms of HF in ATTR-ACT. On top of GDMT, exercise training (ET) remains largely uninvestigated in AC. ET consists of a multidisciplinary approach, including a medical evaluation with modification of cardiovascular risk factors, prescription of a physical exercise program and psychosocial evaluation and is currently recommended with the highest degree of recommendation (in class I, type A level) in current guidelines on HF. To date, there are no data about the efficacy and safety of ET in AC, specifically in the ATTRwt-AC. We hereby present the outlines and the study protocol of the Exercise Rehabilitation and training in Cardiac Amyloidosis (ERICA) study, whose aim is to investigate and analyze the safety and the efficacy of cardiac rehabilitation on patients with AC, specifically those affected by the ATTR-wt form. The present study aims to investigate and analyze, through an interventional longitudinal, controlled, randomized, design, the effects of a structured program of Exercise training in patients with ATTRwt-AC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Established ATTRwt diagnosis
* Heart Failure diagnosis
* Informed consent according to Italian regulations

Exclusion Criteria:

* Unstable Angina
* Acutely decompensated Heart Failure within 1 month before enrollment
* Occurrence of complex ventricular arrhythmias
* Presence of intracavitary thrombus
* recent (< 1 year) thrombophlebitis with or without pulmonary embolism
* Severe obstructive cardiomyopathies
* Severe or symptomatic aortic stenosis
* Uncontrolled inflammatory or infectious diseases
* Any musculoskeletal conditions preventing physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
distance obtained at the 6-minute walk test (6MWD) | Baseline and after 12-weeks of treatment
  distance (meters) obtained at the 6-minute walk test (6MWD) performed at baseline and after 12-weeks of treatment treatment in pooled ET-1 and ET-2 groups compared to No-ET.

SECONDARY OUTCOMES:
N terminal pro brain natriuretic peptide (NT-pro BNP) serum levels | Baseline and after 12-weeks of treatment
  serum levels (ng/ml)
Troponin serum levels | Baseline and after 12-weeks of treatment
  serum levels (ng/ml)
Galectin-3 serum levels | Baseline and after 12-weeks of treatment
  serum levels (ng/ml)
Transthyretin serum levels | Baseline and after 12-weeks of treatment
  serum levels (ng/ml)
Quality of life assessment | Baseline and after 12-weeks of treatment
  Kansas City Questionnaire (ranges 0 to 100 where 100 is the better quality of life score )
Left ventricular ejection fraction (LVEF) | Baseline and after 12-weeks of treatment
  assessed at echocardiography (%)
Left atrial (LA,ml) volume | Baseline and after 12-weeks of treatment
  assessed at echocardiography in ml
global longitudinal strain (GLS) | Baseline and after 12-weeks of treatment
  assessed at echocardiography in %
Tricuspid Annular Plane Systolic Excursion (TAPSE) | Baseline and after 12-weeks of treatment
  assessed at echocardiography in mm
estimated systolic Pulmonary arterial pressure | Baseline and after 12-weeks of treatment
  assessed at echocardiography in mmHg
Right Ventricular Free-wall Strain (RVFWS) | Baseline and after 12-weeks of treatment
  assessed at echocardiography in %
Myocardial work | Baseline and after 12-weeks of treatment
  assessed at echocardiography in mm Hg%
Peak oxygen consumption (VO2 peak) | Baseline and after 12-weeks of treatment
  assessed during Cardiopulmonary exercise test in mL/(kg·min)
Work (Watt) | Baseline and after 12-weeks of treatment
  assessed during Cardiopulmonary exercise test in watt
Respiratory efficiency | Baseline and after 12-weeks of treatment
  minute ventilation (VE)/ carbon dioxide (VCO2) slope assessed during Cardiopulmonary exercise test in watt
Adverse Events | Baseline and after 12-weeks of treatment
  Any adverse Event with special focus on Serious Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M. Marrra, Md,PhD, Principal Investigator — Department of Translational Medical Sciences
Locations (1):
- Department of Translational Medical Sciences, Naples, Italy

IPD SHARING:
Plan to Share IPD: No